CLINICAL TRIAL: NCT06835582
Title: Assessing Concentrations of Methadone and Its Metabolites
Status: Enrolling by invitation | Type: Observational
Sponsor: Cari Health Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB004
Record Dates: First submitted 2025-02-11; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder; Pain
Keywords: Pharmacokinetics; dose curve; electrochemistry; dose taken sensor; personalized dosing; pharmacogenomics
MeSH Terms: conditions — Opioid-Related Disorders; Pain | interventions — Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Methadone — Comparing methadone point of care test to LC-MS to evalutate methadone and its metabolite levels pre dosing and after dosing using the patient's current methadone prescription.

SUMMARY:
An observational proof of concept method comparison study. Comparing Liquid Chromatography -Mass Spectroscopy to a new Quantitative Lateral Flow Immunoassay with an Optical Reader.

DETAILED DESCRIPTION:
CARI Health, Inc.'s long-term goal is to address the problem of high dropout rates of patients receiving medication for opioid use disorder (MOUD; e.g., methadone) treatments, which has increased with the prevalence of fentanyl use, with an innovative point-of-care (PoC) device to enable science-based personalized dosing for patients receiving methadone treatment for opioid use disorder (OUD). The proposed solution consists of a customized analysis device that incorporates proprietary methadone detection technology for quickly measuring methadone and metabolite levels in the blood and calculating the methadone/metabolite ratio (MMR).

To accomplish this long-term goal, the investigators aim to first quantitatively measure methadone doses taken and ethylidene-dimethyl-diphenyl pyrrolidine (EDDP) detection using lateral flow assays. At this stage, the investigators are not testing a device. They are first assessing whether methadone metabolism can be evaluated using lateral flow assays, which are simple paper-based diagnostic strips. The tests work similarly to a home pregnancy test, where a sample (like blood, urine, or saliva) flows along a test strip and interacts with antibodies or other molecules that capture the target substance. No clinical decisions will be made, no treatment will be applied, and no dosing will be changed based on the results learned in this study.

ELIGIBILITY:
Inclusion Criteria:

Age 18-70. A prescription for methadone at a dose of 10mg or more for at least 7 days. Participants may be taking the methadone to treat an OUD or for pain. Taking methadone as prescribed during the last 4 days before consent to participate in the study.

Has been prescribed at least 1 day of take-home doses.

Exclusion criteria for methadone group includes:

Age <18 or >70. A condition preventing or complicating blood collection. Conditions may include dermatological (skin) condition, bleeding diathesis, immunodeficiency, recent blood donation, anemia, end stage renal disease, liver cirrhosis, cancer, congestive heart failure, bleeding diathesis, tuberculosis (TB), active severe depression (e.g., suicidal ideation), or mania symptoms.

Tattoo or piercing close to sampling area. Under a conservatorship.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pain or opioid use disorder that are taking methadone daily.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of whole blood methadone levels with Lateral Flow Assay | 1 day
  whole blood measurement of methadone
Measurement of whole blood methadone metabolite Levels with Lateral Flow Assay | 1 day
  Whole blood measurement of methadone metabolite
Measurement of plasma methadone with LC-MS | 1 day
  plasma methadone with LC-MS
Measurement of plasma methadone metabolite with LC-MS | 1 day
  plasma methadone metabolite with LC-MS

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Semenluk, MD, MD, Principal Investigator — Synergy Research
Locations (1):
- Synergy, Lemon Grove, California, United States

IPD SHARING:
Plan to Share IPD: No